CLINICAL TRIAL: NCT03186898
Title: A Phase III Randomized Trial of Protons Versus Photons for Hepatocellular Carcinoma
Brief Title: Radiation Therapy With Protons or Photons in Treating Patients With Liver Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GI003; NCI-2016-02009 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GI003 (Other: NRG Oncology); NRG-GI003 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v7; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (proton therapy) (Experimental): Patients undergo proton therapy over 15-24 days for 5 or 15 fractions. Patients undergo CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy
- Arm II (photon therapy) (Experimental): Patients undergo photon therapy over 15-24 days for 5 or 15 fractions. Patients undergo CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo proton therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm I (proton therapy)
Radiation: Radiation Therapy — Undergo photon therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm II (photon therapy)

SUMMARY:
This phase III trial studies how well radiation therapy with protons works compared with photons in treating patients with liver cancer. Radiation therapy, such as photon therapy, uses high energy x-rays to send the radiation inside the body to the tumor while proton therapy uses a beam of proton particles. Proton therapy can stop shortly after penetrating through the tumor and may cause less damage to the surrounding healthy organs and result in better survival in patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if overall survival (OS) is different for hepatocellular carcinoma patients treated with protons compared to photons.

SECONDARY OBJECTIVES:

I. To determine the difference in progression-free-survival (PFS) in patients with hepatocellular carcinoma (HCC) treated with protons compared to patients with HCC treated with photons.

II. To determine the difference in local progression (LP) in patients with HCC treated with protons compared to patients with HCC treated with photons.

III. To determine differences in toxicity in patients with HCC treated with protons versus photons.

IV. To determine differences in fatigue, as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) fatigue in patients with HCC treated with protons, versus photons; as well as quality-adjusted survival, if the primary endpoint is met.

V. To determine if there are correlations between the baseline values of hepatocyte growth factor (HGF) and outcomes (OS/PFS/fatigue).

EXPLORATORY OBJECTIVES:

I. To determine differences in overall quality of life, measured by Functional Assessment of Cancer Therapy-Hepatobiliary Cancer (FACT-Hep) in patients with HCC treated with protons.

II. Biospecimen collection for future correlative science projects.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo proton therapy over 15-24 days for 5 or 15 fractions.

ARM II: Patients undergo photon therapy over 15-24 days for 5 or 15 fractions.

Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) or radiographically-proven (based on the American Association for the Study of Liver Diseases [AALSD] criteria) unresectable or locally recurrent hepatocellular cancer prior to registration
* Appropriate stage for study entry based on the following diagnostic workup:

  * All patients must have computed tomography (CT) scan chest/abdomen/pelvis with multiphasic liver CT scan prior to registration; if CT contrast is contraindicated, CT chest without contrast and magnetic resonance imaging (MRI) of abdomen is permitted
  * Participants must have measurable disease at study entry, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 2 cm with conventional techniques or as > 1 cm with spiral CT scan
  * Patient must have 3 or fewer single or multinodular tumors; for patients with a single lesion, lesion must be 15 cm or less in greatest dimension; for patients with two lesions, no lesion may be greater than 10 cm in greatest dimension; for patients with three lesions, no lesion may be greater than 6 cm in greatest dimension; portal vein involvement or thrombosis combined with a single lesion that is >= 1 cm and =< 15 cm in greatest dimension is allowed
* Age >= 18
* Zubrod performance status 0-1 within 30 days prior to registration
* Negative urine or serum pregnancy test for women of childbearing potential within 7 days prior to study entry
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3
* Platelets >= 50,000 cells/mm^3
* Hemoglobin >= 9.0 g/dl; (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 9.0 g/dl is acceptable)
* Total bilirubin < 4 x institutional upper limit of normal (ULN)
* Transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) < 6 x institutional ULN
* Albumin >= 2.5 g/dl
* Creatinine < 2 mg/dl
* Prior chemotherapy, targeted biological therapy (e.g. sorafenib), surgery, transarterial chemoembolization (TACE), ablation for present disease is acceptable
* Must have Child-Turcotte-Pugh (CTP) A or B7
* The patient or a legally authorized representative must provide study-specific informed consent prior to study registration

Exclusion Criteria:

* PRIOR TO STEP ONE REGISTRATION:
* Definitive clinical or radiologic documentation of extrahepatic tumor, defined as extrahepatic metastases or malignant nodes (that enhance with typical features of HCC) > 3.0 cm, in sum of maximal diameters (e.g. presence of one 3.4 cm metastatic lymph node or two 2 cm lung lesions); note that benign non-enhancing periportal lymphadenopathy is not unusual in the presence of hepatitis and is permitted, even if the sum of enlarged nodes is > 2.0 cm
* Uncontrolled prior invasive malignancy, excluding the current diagnosis
* Systemic chemotherapy for the study cancer < 2 weeks prior to registration
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* HIV positive with CD4 count < 200 cells/microliter; note that patients who are human immunodeficiency virus (HIV) positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter prior to registration; note also that HIV testing is not required for eligibility for this protocol; this exclusion criterion is necessary because the treatments involved in this protocol may be significantly immunosuppressive
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields (to include Y90)
* Prior liver transplant
* PRIOR TO STEP TWO RANDOMIZATION:
* Unable to obtain confirmation of payment coverage (insurance or other) for either possible treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-01-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death due to any cause assessed up to 4 years
  Will be estimated by the Kaplan-Meier method. The distributions of OS between treatment arms will be compared using the log rank test. The final analysis will occur after at least 125 deaths have occurred and will include: tabulation of all cases entered and those excluded from the analyses with the reasons for exclusion, distributions of important prognostic baseline variables, the frequencies and severity of adverse events by treatment arm, treatment delivery compliance, observed results with respect to the primary endpoint of OS. Will be tested with a 2-sided significance level of 0.049.
Treatment effect | Up to 4 years
  Will be performed using the Cox proportional hazard regression model.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization to the date of first PFS failure or last follow-up for patients without a reported PFS event assessed up to 4 years
  Will be estimated by the Kaplan-Meier method and compared using the log rank test. The Cox proportional hazard regression model will be used.
Local progression (LP) | From the date of randomization to the date of first LP or date of last follow-up for patients without an LP event reported assessed up to 4 years
  Will be estimated by the cumulative incidence method and compared using Gray's test. The Fine-Gray regression model will be used to analyze.
Incidence of adverse events | Up to 4 years
  Will be assessed by Common Terminology Criteria for Adverse Events version 4. A Chi-square test will be used to compare the number of patients with at least 1 grade 3 or higher adverse events between the treatment arms.
Fatigue | Baseline up to 6 months
  Will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) fatigue short form version 1.0 8a.
Change in fatigue | Baseline up to 1 month
  Will be compared between treatment arms using a t-test. If the data do not satisfy the normality assumption, a Wilcoxon test may be used instead.
Quality-adjusted survival | Baseline up to 12 months
  Will be evaluated and compared using European Quality of Life Five Dimension Three Level Questionnaire (EuroQol 5D).
Plasma hepatocyte growth factor (HGF) levels | At baseline
  Will be dichotomized at the median value and evaluated for prognostic significance using Cox regression model at a 2-sided significance level of 0.05. Additionally, predictive analyses will be done by treatment arm and an exploratory test of HGF by treatment interaction, with the understanding that there will be reduced power for the predictive analyses under the same effect size assumptions. However, there may be sufficient power if there is large interaction.

OTHER OUTCOMES:
Overall quality of life by Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) version 4 | Baseline up to 12 months
  Differences between treatment arms in the overall score, the four domains (physical, social, emotional, and functional well-being), and the additional concerns subscale will also be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S Hong, Principal Investigator — NRG Oncology
Locations (27):
- United States (27):
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - New York Proton Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington

REFERENCES:
- [Derived] Duda DG. Targeting Tumor Microenvironment in Liver Cancers: Rationale, Current Progress, and Future Perspective. Keio J Med. 2022;71(3):71. doi: 10.2302/kjm.71-004-ABST. PMID 36155490